CLINICAL TRIAL: NCT03995199
Title: A Comparison of Speech Outcome in Pediatric Cleft Patients, After Modified Furlow Palatoplasty in Combination With Intravelar Veloplasty According to Sommerlad, or Modified Furlow Palatoplasty Alone
Brief Title: A Comparison of Speech Outcome in Pediatric Cleft Patients, After Modified Furlow-Sommerlad Palatoplasty in Comparison to Modified Furlow Palatoplasty Alone
Acronym: SPEAC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: AZ Sint-Jan AV (Other)
Responsible Party: Principal Investigator, Krisztian Nagy, principal investigator, maxillofacial surgeon, AZ Sint-Jan AV
Other Study IDs: B049201629483
Record Dates: First submitted 2019-06-19; First posted 2019-06-21 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-02

CONDITIONS: Cleft Palate Children
Keywords: speech evaluation; modified Furlow palatoplasty; Sommerlad intravelar veloplasty

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Furlow group: All cleft palate patients surgically treated with a modified Furlow technique since January 2012
- Furlow + Sommerlad group: All cleft palate patients surgically treated with a modified Furlow technique in combination with an intravelar veloplasty by Sommerlad

SUMMARY:
Nowadays, surgical success of cleft palate patients is ascribed to the sufficiency of velopharyngeal closure, and the associated speech results such as voice nasality, resonance and articulation. The investigators aim to evaluate if the surgical modified Furlow palatoplasty in combination with the intravelar veloplasty according to Sommerlad significantly reduces the number of pediatric patients with abnormal speech between five and seven years of age, as measured with the four-point scale recently published by Nguyen et al.(2015), in comparison to the conventional modified Furlow technique.

study design A prospective cohort trial. All cleft palate patients surgically treated with a modified Furlow technique since January 2012 or a modified Furlow technique in combination with an intravelar veloplasty by Sommerlad routinely undergo an annual speech evaluation by the speech language pathologist of the cleft team. At the age of five, eligible patients that are in continuous follow-up by the cleft team at our hospital, will be asked for consent to register their demographic, surgical and speech-related data. In addition, the parents of cleft patients will be asked to complete a quality of life questionnaire concerning their child, at the time of speech evaluation through self-report or through an interview with the clinical research coordinator.

The investigators hypothesise that the combined modified Furlow and Sommerlad palatoplasty leads to a minimal 50% reduction in the proportion of children with abnormal speech, as defined by the four-point scale recently published by Nguyen et al.(2015), compared to patients that underwent a Modified Furlow technique alone.

conclusion Although the technique by Sommerlad has shown promising results, prospective trials comparing postoperative speech outcome after different surgical techniques, are lacking. The present trial could offer objective results to validate the current surgical treatment protocol implemented at our department.

DETAILED DESCRIPTION:
Nowadays, surgical success of cleft palate patients is ascribed to the sufficiency of velopharyngeal closure, and the associated speech results such as voice nasality, resonance and articulation. The investigators aim to evaluate if the surgical modified Furlow palatoplasty in combination with the intravelar veloplasty according to Sommerlad significantly reduces the number of pediatric patients with abnormal speech between five and seven years of age, as measured with the four-point scale recently published by Nguyen et al.(2015), in comparison to the conventional modified Furlow technique.

study design A prospective cohort trial. All cleft palate patients surgically treated with a modified Furlow technique since January 2012 or a modified Furlow technique in combination with an intravelar veloplasty by Sommerlad routinely undergo an annual speech evaluation by the speech language pathologist of the cleft team. At the age of five, eligible patients that are in continuous follow-up by the cleft team at our hospital, will be asked for consent to register their demographic, surgical and speech-related data. In addition, the parents of cleft patients will be asked to complete a quality of life questionnaire concerning their child, at the time of speech evaluation through self-report or through an interview with the clinical research coordinator.

The investigators hypothesise that the combined modified Furlow and Sommerlad palatoplasty leads to a minimal 50% reduction in the proportion of children with abnormal speech, as defined by the four-point scale recently published by Nguyen et al.(2015), compared to patients that underwent a Modified Furlow technique alone.

conclusion Although the technique by Sommerlad has shown promising results, prospective trials comparing postoperative speech outcome after different surgical techniques, are lacking. The present trial could offer objective results to validate the current surgical treatment protocol implemented at our department.

ELIGIBILITY:
Inclusion Criteria:

* Patients should have a clinically diagnosed cleft of the hard and/or soft palatum, with or without involvement of the lip or nose (Veau classification I to IV (see Appendix 1).
* Patients should have undergone a modified Furlow palatoplasty or modified Furlow according to Sommerlad in the AZ Sint-Jan Brugge-Oostende av
* Patients should receive their postoperative care and speech therapy by the cleft team of the general hospital Sint-Jan Bruges
* Patients should be in the fifth life year at time of speech evaluation
* Patients should be Dutch-speaking as a maternal language

Exclusion Criteria:

* Patients not meeting the abovementioned inclusion criteria
* Patients that received a corrective surgical procedure for velopharyngeal dysfunction after the modified Furlow technique alone, or in combination with the intravelar veloplasty by Sommerlad
* Patients that are bi- or multilingual
* Patients with clinically diagnosed mild hearing difficulties (i.e. ASHA classification: hearing loss >25dB)30
* Patients with a clinically diagnosed stutter
* Patients with clinically diagnosed cognitive and/or motoric disabilities
* Patients that received intensive speech therapy prior to their fifth life year can be included, but will be analyzed separately(subgroup analysis)
* Note: The number of patients with a uni- or bilateral cleft involving the lip or nose should be comparable between both groups, since this can interfere with speech and could bias comparison of speech outcome between different cleft subgroups.

Ages: 5 Years to 7 Years | Sex: All
Age Groups: Child
Study Population: Patients with a clinically diagnosed cleft of the hard and/or soft palatum, that are treated surgically with a modified Furlow palatoplasty or a modified Furlow palatoplasty in combination with an intravelar veloplasty by Sommerlad. Patients should receive their postoperative care and annual speech evaluation by the cleft team of the AZ Sint-Jan Brugge-Oostende av.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2017-09-13 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
proportion of children with abnormal speech, as defined by the four-point scale recently published by Nguyen et al.(2015) | at time of routine speech evaluation between age 5-7 years old
  proportion of children with abnormal speech, as defined by the four-point scale recently published by Nguyen et al.(2015)

SECONDARY OUTCOMES:
prevalence of speech problems, as defined by the perceptual evaluation | at time of routine speech evaluation between age 5-7 years old
  prevalence of speech problems, as defined by the perceptual evaluation
prevalence of speech problems, as defined by the objective speech evaluation (nasometry) | at time of routine speech evaluation between age 5-7 years old
  prevalence of speech problems, as defined by the objective speech evaluation (nasometry)
incidence of 30-day postoperative complications | within 30 days postoperative
  incidence of 30-day postoperative complications
PVRQOL questionnaire, as a measure of quality of life | at time of routine speech evaluation between age 5-7 years old
  PVRQOL questionnaire, as a measure of quality of life
COHIP questionnaire, as a measure of quality of life | at time of routine speech evaluation between age 5-7 years old
  COHIP questionnaire, as a measure of quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- Division of oral and maxillofacial surgery, Department of Surgery, AZ Sint-Jan Brugge-Oostende AV, Bruges, Belgium

IPD SHARING:
Plan to Share IPD: No